CLINICAL TRIAL: NCT06333977
Title: A First in Human, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LC542019 in Healthy Subjects and Subjects With T2DM
Brief Title: A Study of LC542019 in Healthy Subjects and Subjects With T2DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: LG-GQCL001
Record Dates: First submitted 2023-07-31; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Healthy; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LC542019 (Experimental): oral dose, once daily.
  Interventions: Drug: LC542019
- Placebo (Placebo Comparator): matching placebo capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LC542019 — oral dose, once daily
  Arms: LC542019
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
to assess the safety, tolerability, Pharmacokinetics and Pharmacodynamics in healthy subjects and subjects with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
The study will be conducted in 2 parts:

Part 1 (Single Ascending Dose) This part will include 6 sequential dose cohorts (S1-S6).

Part 2 (Multiple Ascending Dose) This part will include 5 sequential dose cohorts (M1-M5). Cohorts M1-M4 will enroll healthy subjects. Cohort M5 will enroll subjects with T2DM.

ELIGIBILITY:
For healthy subjects:

Inclusion criteria

* Adults ≥ 18 to ≤ 55 years.
* Body mass index (BMI) ≥18.5 to ≤ 30.0 kg/m2
* Female subjects must be non-pregnant and non-lactating. Females of childbearing potential must use at least two of the medically accepted contraceptive methods, table at least 4 weeks prior to the screening.
* Ability to provide written informed consent.

Exclusion Criteria

* History of or current diagnosis of Diabetes Mellitus Type 1 or Diabetes Mellitus Type 2
* History of or current significant diagnosis of cardiovascular, respiratory, hepatic, renal, gastrointestinal endocrine, hematological, or neurological disorders or abnormalities, or other major systemic disease
* History of or presence of clinically significant ECG findings
* History of or acute significant gastrointestinal disorder

For T2DM subjects:

Inclusion criteria

* Adults ≥ 18 to ≤ 70 years.
* Body mass index (BMI) ≥18.5 to ≤ 35.0 kg/m2 with stable body weight by history for 3 months
* Subjects with T2DM > 6 months, on stable therapy with metformin monotherapy.
* Female subjects must be non-pregnant and non-lactating. Females of childbearing potential must use at least two of the medically accepted contraceptive methods, table at least 4 weeks prior to the screening.
* Ability to provide written informed consent.

Exclusion Criteria

* History of or current diagnosis of Diabetes Mellitus Type 1
* A subject who has acute proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, especially autonomic neuropathy
* Recurrent major hypoglycemia or hypoglycemic unawareness or recent ketoacidosis
* Current use of any prescribed or non-prescribed drugs (other than current treatment for diabetes mellitus or birth control methods)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Incidence, severity of adverse events | up to 4 weeks

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) in Plasma | up to 4 weeks
Renal Clearance (CLR) in urine | up to 2 weeks

OTHER OUTCOMES:
Cardiodynamic evaluation | up to 4 weeks
  concentration-QTc analysis
Fasting Plasma Glucose | up to 4 weeks
HbA1c | up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP (PPD Clinical Research Unit, Las Vegas), Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No